CLINICAL TRIAL: NCT07328191
Title: Quality of Life-based Transfusion in Refractory MDS or AML Under Advanced Palliative Care and Supportive Treatment.
Brief Title: Quality of Life-Guided Transfusion in Refractory MDS or AML
Acronym: Q-TRANS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-AOI-02
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: MDS; AML, Adult; Anemia
Keywords: palliative care; Chronic Transfusion-Dependent Anemia; Transfusion-dependent anemia; MDS; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to one of two parallel groups: a standard hemoglobin-based red blood cell transfusion strategy or a quality-of-life-guided transfusion strategy based on EQ-5D-5L assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemoglobin-Based Transfusion Strategy (No Intervention): Red blood cell transfusions are performed according to standard hemoglobin thresholds (Hb <7 g/dL, or <8 g/dL in patients with cardiovascular comorbidities). Standard of care arm
- Quality of Life-Guided Transfusion Strategy (Experimental): Red blood cell transfusions are performed when a clinically significant deterioration (≥1 level decrease in at least one EQ-5D-5L domain compared to baseline) is observed
  Interventions: Other: Red blood cell transfusions based on EQ-5D-5L questionnaire

INTERVENTIONS:
Other: Red blood cell transfusions based on EQ-5D-5L questionnaire — Red blood cell transfusions are administered based on patient-reported quality-of-life assessments using the EQ-5D-5L questionnaire, collected weekly. A transfusion is performed when a deterioration of at least one level in any EQ-5D-5L dimension is observed.
  Arms: Quality of Life-Guided Transfusion Strategy

SUMMARY:
Patients with refractory myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML) in exclusive palliative care frequently receive red blood cell transfusions based on hemoglobin thresholds, despite limited evidence of clinical benefit in this setting.

This prospective randomized study compares a standard hemoglobin-based transfusion strategy to a quality-of-life-guided strategy using the EQ-5D-5L questionnaire, with the aim of reducing transfusion burden while maintaining patient safety and quality of life.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized interventional study conducted in patients with transfusion-dependent refractory MDS or AML receiving exclusive palliative care. Palliative Care

Patients are randomized to either a standard transfusion strategy based on hemoglobin thresholds or a quality-of-life-guided strategy in which red blood cell transfusions are triggered by a clinically significant deterioration in EQ-5D-5L score.

The study aims to evaluate whether a quality-of-life-guided transfusion strategy can safely reduce the number of red blood cell transfusions without negatively impacting patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Diagnosis of refractory MDS or AML, receiving palliative care only.
* Anaemia with haemoglobin ≤ 8 g/dl at inclusion (or ≤ 9 g/dl if associated with cardiovascular disease).
* Transfusion dependency, defined as requiring more than 2 GR transfusions every 8 weeks.
* No vitamin B9, vitamin B12 or iron deficiency.
* Ability to understand and sign the informed consent form.
* Ability to comply with the schedule of visits and other protocol requirements.

Non inclusion Criteria:

* Previous malignant disease other than MDS or AML (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast).
* Active uncontrolled infection (hepatitis B or C, HIV).
* Use of G-CSF.
* Confirmed neurocognitive disorders (based on prior diagnosis or clinical assessment by the investigator) impairing comprehension, consent or the ability to reliably complete the EQ-5D-5L questionnaire.
* Active uncontrolled heart disease.
* Active haemolytic anaemia.
* Recent major surgery.
* Life-threatening complications of MDS/AML.
* Presence of another serious or unstable disease which, in the investigators' opinion, would make participation in the study inappropriate or risky for the patient's safety.
* Vulnerable individuals.

Exclusion Criteria:

* Immediate severe complications related to MDS/AML, such as uncontrolled bleeding, pneumonia with hypoxia or shock, or severe disseminated intravascular coagulopathy.
* Withdrawal of the patient's voluntary informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02-09 (Actual); Primary Completion 2027-02-09 (Estimated); Study Completion 2028-02-09 (Estimated)

PRIMARY OUTCOMES:
Number of Red Blood Cell Transfusions | 2 months
  Total number of red blood cell units transfused during the 2-month follow-up period.

SECONDARY OUTCOMES:
Quality of Life (EQ-5D-5L) | from baseline to 1 month and 2 months.
  Change in quality-of-life scores
Overall Survival | from inclusion to 2 months
  Survival status

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cluzeau, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No